CLINICAL TRIAL: NCT07080944
Title: Sentinel Lymph Node Biopsy After Neoadjuvant Chemotherapy in Inflammatory Breast Cancer: a Prospective Trial
Brief Title: Sentinel Lymph Node Biopsy After Neoadjuvant Chemotherapy in IBC
Acronym: SYMPHONY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UID 4964; L2-371 (Other: Comitato Etico Territoriale Lombardia 2)
Record Dates: First submitted 2025-07-15; First posted 2025-07-23 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Invasive Breast Carcinoma; Sentinel Lymph Node Biopsy (SLNB); Neoadjuvant Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Patients with SLN visualization.
  Interventions: Procedure: SLN identification using technetium-99m
- Group 2a (Experimental): Patients with no pre-surgery SLN visualization and intra-surgery SLN identification.
  Interventions: Procedure: SLN intra-operatory identification with radioguided surgery
- Group 2b (Active Comparator): Patients with no pre-surgery SLN visualization and no intra-surgery SLN identification.
  Interventions: Procedure: Axillary Limph Node Dissection (ALND)

INTERVENTIONS:
Procedure: SLN identification using technetium-99m — SLN Biopsy after pre-surgery positive SLN visualization.
  Arms: Group 1
Procedure: SLN intra-operatory identification with radioguided surgery — SLN biopsy after no pre-surgery SLN visualization using technetium-99m and intra-surgery SLN identification.
  Arms: Group 2a
Procedure: Axillary Limph Node Dissection (ALND) — Axillary Limph Node Dissection (ALND) after no pre-surgery SLN visualization using technetium-99m and no intra-surgery SLN identification.
  Arms: Group 2b

SUMMARY:
This study will prospectively determine the feasibility and oncological safety of sentinel lymph node biopsy (SLNB) after neoadjuvant chemotherapy (NACT) in inflammatory breast cancer patients traditionally considered ineligible for SLNB due to locally advanced cancer with skin/chest wall involvement (cT4d) and heavy nodal burden at presentation (cN1/N2). This study will also assess the identification rate of sentinel lymph-node (SLN) (using single tracer mapping) after NACT in this patient population. Finally, the study will determine the long-term outcome of such cohort.

ELIGIBILITY:
Inclusion Criteria:

* Female patients over 18 years of age with clinically and biopsy-proven stage IIIB cT4d cN0-2 M0 breast cancer as assessed by clinical exam and imaging
* Patients receiving NACT and having a nodal complete clinical response (ycN0) as assessed by physical exam and imaging (ultrasound and PET)
* Ability to understand and willingness to sign informed consent document and comply with study procedures

Exclusion Criteria:

* Patients with cN3 stage at diagnosis
* Participants with stage IV (metastatic) breast cancer
* Participants with positive contralateral axillary nodes identified on standard imaging studies (mammograpy, MRI, ultrasound) and cito-histologically ascertained
* Patients with a prior history of ipsilateral breast cancer
* Pregnant patients
* Patients after NACT with persistent palpable axillary nodes, as assessed by physical exam, or with persistent pathological axillary nodes, as assessed by imaging
* Patients not consenting to ALND

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-12-12 (Actual); Primary Completion 2030-07 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
intraoperative SLN identification rate. | 3 Months
  Evaluation of the feasibility of SLNB in a selected cohort of IBC patients operated who responded to systemic NACT in the axillary nodes, achieving complete clinical response (ycN0). The feasibility of SLNB, defined as the intraoperative SLN identification rate, will be calculated as the proportion of patients with successfully identified intraoperative SLNs among the enrolled patients.

SECONDARY OUTCOMES:
Disease-free survival (DFS) | 5 years.
  DFS will be defined as the time from surgery to loco-regional recurrence, metastasis, other primary non-breast carcinomas, or death, whichever occurs first.
Distant recurrence-free survival (DRFS) | 5 years
  DRFS will be defined as the time from surgery to distant recurrence or death from any cause, whichever occurs first.
Breast cancer-specific survival (BCSS) | 5 years
  BCSS will be defined as the time from surgery to death due to breast cancer.
Overall survival (OS) | 5 years
  OS will be defined as the time from surgery to death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- European Institute of Oncology, Milan, Italy